CLINICAL TRIAL: NCT03275168
Title: Developing a Dyadic Intervention for STI/HIV Prevention in Youth
Brief Title: Developing a Dyadic Intervention for Sexually Transmitted Infection (STI)/HIV Prevention in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00148707; 1R21HD090498-01A1 (NIH)
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Exposure to Sexually Transmissible Disorder (Event)
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants will receive individual evidence-based STI/HIV prevention intervention (Sister to Sister Teen for female participants and Focus on the Future for male participants) for STI prevention
  Interventions: Behavioral: Individual evidence-based STI/HIV prevention intervention
- Intervention (Experimental): Participants will receive individual evidence-based STI/HIV prevention intervention (Sister to Sister Teen for female participants and Focus on the Future for male participants) for STI prevention plus dyadic counseling and negotiation practice with partner
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Sexual partners will receive dyadic counseling and support for condom negotiation after receipt of individual evidence based HIV/STI prevention intervention (Sister-to-Sister (female) and Focus on the Future (male).
  Arms: Intervention
Behavioral: Individual evidence-based STI/HIV prevention intervention — Sexual partners will receive individual evidence-based HIV/STI prevention counseling without partner debrief and/or practice negotiating condom use.
  Other Names: Sister to Sister / Focus on the Future
  Arms: Control

SUMMARY:
This pilot project will evaluate the feasibility, acceptability, and preliminary effectiveness of a couples-based behavioral intervention [COUPLES] that augments individual evidence-based interventions with joint health education counseling for STI-affected AYA dyads within a primary care setting.

DETAILED DESCRIPTION:
While public health programs have demonstrated modest success in reducing the adolescent and young adult (AYA) risk for STI/HIV, significant health disparities remain. The risk of STI/HIV is not uniform among AYA. AYA residing in segregated urban communities with high STI prevalence and complicated sexual networks face even greater risk for disease and associated complications. Additional supports designed to increase engagement in care and reduce STI acquisition and transmissions are urgently needed to meet the sexual health and reproductive health goals for the nation. Overwhelmingly, AYA STI prevention interventions have targeted individuals and individual-level factors. While effective, these interventions do not adequately address other important influences affecting AYA risk for STI/HIV, such as partner or relationship influences on sexual decision-making and behavior. Partner notification and treatment is a key strategy for disease control and has previously been tested among adults for STI/HIV prevention work but has yet to be evaluated for AYA. Our prior research demonstrates that AYAs with complicated STIs are likely to notify their partners to seek treatment (88-92%); however, AYAs receiving brief behavioral interventions, relative to those receiving standard of care were 3 times more likely to be successful in arranging for their partner's treatment. Thus, partner interventions may hold promise for harnessing the power of relationship dynamics to enhance sexual decision-making, communication, and subsequent health behaviors. The investigators propose to pilot test an intervention designed to change sexual health outcomes by understanding partners and the learning environment related to sex [COUPLES] by simultaneously delivering two evidence-based STI/HIV prevention interventions Sister-to-Sister Teen and Focus on the Future. The simultaneous delivery of effective interventions will be augmented with a joint partner health education counseling session focused on enhancing communication and negotiation of safe sexual practices within the relationship. If successful, this pilot will support the development of a larger trial designed to evaluate the effectiveness of this approach in the busy primary care setting by providing evidence that AYA can and will safely engage their partners in a supportive primary care setting that integrates high quality treatment with evidence-based STI/HIV prevention interventions delivered by health educator teams.

ELIGIBILITY:
Inclusion Criteria:

The index patient must be

* 16-25 years
* Engage in male-female [heterosexual] intercourse
* Permanently reside in the Greater Baltimore Metropolitan Area (GBMA)
* Willing to recruit their main sexual partner for the study
* Willing to participate in a single individual session with a health educator followed by a joint debriefing session together
* Willing to be contacted in 6-8 weeks for a telephone interview

The partner must be

* 16-30 years
* Engage in male-female [heterosexual] intercourse with the index patient
* Permanently reside in the greater Baltimore Metropolitan Area
* Willing to participate in a single individual session with a health educator followed by a joint debriefing session together
* Willing to be contacted in 6-8 weeks for a telephone interview

Exclusion Criteria:

* Index participants and partners who are unable to communicate with staff or participate in study procedures due to cognitive, mental, or language difficulties will not be eligible for recruitment into the study.
* Dyads will also be excluded if in same-sex main partnership or a member of the couple is currently enrolled in another sexual behavior study, one or both partners has a known concurrent HIV infection, one or more partners has a pending incarceration, there is more than five years age difference between the two partners and one partner is <16 years of age, or there is evidence of intimate partner violence (IPV) in the relationship.
* Individuals who screen positive for IPV will be referred to local resources for assistance.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Heterosexual dyads based on female and male biology recruited for study.
Enrollment: 68 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Trent, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot trial. De-identified data will be presented in aggregate in professional presentations and publications.

REFERENCES:
- [Derived] Trent M, Yusuf HE, Rowell J, Toppins J, Woods C, Huettner S, Robinson C, Fields EL, Marcell AV, DiClemente R, Matson P. Dyadic Intervention for Sexually Transmitted Infection Prevention in Urban Adolescents and Young Adults (The SEXPERIENCE Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 May 25;11(5):e29389. doi: 10.2196/29389. PMID 35612881

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 participants were eligible for enrollment in the control arm and 45 participants were eligible for enrollment in the intervention arm. However, 34 in the control arm and 34 in the intervention arm (of the total eligible subjects) returned to be enrolled in the study.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 34 | 34
Completed | 27 | 25
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 1 | 7
  Between 18 and 65 years | 28 | 33 | 61
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (2.6) | 23.5 (2.4) | 22.3 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 18 | 17 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 34 | 68
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by the Number of Participants Who Are Enrolled With a Partner
Description: Recruitment (as a measure of feasibility) will be assessed by calculating the number of eligible patients who return with a partner to the study appointment and consent to participate in the study.
Time Frame: 24 months
Population: The population for analysis is the number of those who were eligible to enroll, not the number who were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 44 | 45
Participants | 17 | 17

2. Secondary Outcome: Acceptability as Assessed by Number of Participants Available for Week 6-8 Interview
Description: Retention for the 6-8 week interview will also be calculated as a measure of acceptability.
Time Frame: 6-8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 34 | 34
Participants | 27 | 25

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT03275168/Prot_SAP_000.pdf